CLINICAL TRIAL: NCT05057949
Title: A Single-center, Open, Self-controlled Design Clinical Study to Evaluate the Pharmacokinetic Effects of Rifampicin or Itraconazole on Single-dose Laolotinib Mesylate Capsules in Healthy Subjects
Brief Title: A Study to Evaluate Drug-Drug Interaction of Larotinib With Itraconazole and Rifampin in Healthy Adult Participants
Acronym: Z650
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Z650-DDI-104
Record Dates: First submitted 2021-08-31; First posted 2021-09-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Rifampin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A, Treatment Sequence(Larotinib-Larotinib/Rifampin) (Experimental): Larotinib , capsules (150mg*2+50mg*1), at Hour 0 on Day 1 followed by an overnight fast. On Days 15 to 26, participants received rifampin 600 mg as capsules, orally, once daily (QD) and Larotinib 350 mg as capsules, orally was coadministered on Day 20. There was a washout period of 13 days between the two treatments.
  Interventions: Drug: Larotinib; Drug: Rifampin
- Part B, Treatment Sequence(Larotinib-Larotinib/itraconazole) (Experimental): Larotinib , capsules (150mg*2+50mg*1), at Hour 0 on Day 1 followed by an overnight fast. On Days 15 to Day 25, participants received itraconazole 200 mg solution, orally, once daily (QD) on Days 15 to Day 25 and a single oral dose of Larotinib 350 mg as capsule was coadministered on Day 19 (Treatment B). There was a washout period of 13 days between the two treatments.
  Interventions: Drug: Larotinib; Drug: Itraconazole

INTERVENTIONS:
Drug: Larotinib — Larotinib Capsules
  Other Names: Z650
Drug: Rifampin — Rifampin Capsules
  Other Names: Rifampin Capsules
  Arms: Part A, Treatment Sequence(Larotinib-Larotinib/Rifampin)
Drug: Itraconazole — Itraconazole Capsules
  Other Names: Itraconazole Capsules
  Arms: Part B, Treatment Sequence(Larotinib-Larotinib/itraconazole)

SUMMARY:
The purpose of this study is to characterize the effect of rifampin (Part A) and itraconazole(Part B) on the single-dose pharmacokinetics (PK) of Larotinib in healthy adult participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called Larotinib (Z650). The study assessed the drug-drug interaction of Larotinib with either a strong cytochrome P-450 (CYP)3A inducer, rifampin (Part A) , or with a strong CYP3A inhibitor itraconazole (Part B) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent was signed before the study, and the content, process and possible adverse reactions of the study were fully understood;
2. Without Plan for pregnancy or pregnant within 6 months from screening to the last dose of the study drug;
3. Healthy, adult, male or female, 18 - 55 years of age;
4. Male subjects should weigh at least 50 kg and female subjects should weigh at least 45 kg. Body mass index (BMI) ≥18.0 and ≤28.0 kg/m2;
5. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs and physical examination.

Exclusion Criteria:

1. Average daily smoking >5 cigarettes in 3 months before the study;
2. Known allergic reactions or hypersensitivity to any excipient of the study drug formulation(s).
3. History of alcoholism(defined as Alcohol consumption of > 14 units/week);
4. Those with positive urine drug screening or those with a history of drug abuse or drug use in the past five years ;
5. Blood donation or significant blood loss (>450 mL) within 3 months prior to screening;
6. Have dysphagia or have gastrointestinal, liver, or kidney disease (whether cured or not) that affects drug absorption or excretion within 6 months prior to screening;
7. Have any medical condition that increases the risk of bleeding, such as hemorrhoids, acute gastritis, or stomach and duodenal ulcers ;
8. Use of any prescription drugs, over-the-counter drugs, any vitamin products or herbal medicines in the 14 days prior to screening;
9. Any drugs that changed the activity of liver drug enzymes, such as barbiturates and rifampicin, were taken within 30 days before screening;
10. Have taken the following inhibitors or inducers of CYP3A4, CYP2C8, CYP2C19 and P-GP within 30 days before screening;
11. Patients who had taken special diet (including pitaya, mango, grapefruit, etc.) or had strenuous exercise, or had other factors affecting drug absorption, distribution, metabolism and excretion, as judged by the researcher, within 14 days before screening ;
12. Participants who have participated in any drug clinical trials within 3 months prior to screening and have used the test drug (subjects may be enrolled in the study if they dropped out of the study prior to dosing, i.e., were not randomized or received dosing) ;
13. Abnormal abdominal ultrasonography, chest radiography, ECG examination is clinically significant, or the corrected QT interval (QTcF) of ECG >470ms during screening period ;
14. Female subjects were lactating or had positive blood pregnancy results at screening or check in;
15. Laboratory examination is abnormal and clinically significant, or the following diseases (including but not limited to gastrointestinal, renal, liver, neurological, hematological, endocrine, tumor, lung, immune, psychiatric or cardiovascular and cerebrovascular diseases) are clinically significant as found within 12 months prior to screening;
16. Viral hepatitis (including hepatitis B and C), HIV antigen/antibody or treponema pallidum antibody was positive at screening;
17. Acute illness or concomitant medication was occurred from the screening to the first administration of the experimental drug;
18. Subjects who consume chocolate, any food or drink containing caffeine or rich in xanthine within 24 hours before taking the study drug;
19. Alcohol breath test is positive at check-in.
20. Subjects who received vaccination within 28 days prior to screening or who plan to receive vaccination during the trial ;
21. The investigator deemed the subject unsuitable for this study for any reason

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 pre-dose at multiple time points (up to 192 hours) post-dose
  Maximum Observed Plasma Concentration of Larotinib
AUC∞ | Day 1 pre-dose at multiple time points (up to 192 hours) post-dose
  Area Under the Plasma Concentration-time Curve from Time 0 to Infinity, calculated using the observed value of the last quantifiable concentration for Larotinib

SECONDARY OUTCOMES:
AUClast | Day 1 pre-dose at multiple time points (up to 192 hours) post-dose
  Area Under the Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration for Larotinib
Tmax | Day 1 pre-dose at multiple time points (up to 192 hours) post-dose
  Time to Reach the Maximum Plasma Concentration (Cmax) for Larotinib

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No